CLINICAL TRIAL: NCT02740270
Title: A Phase I/Ib Open-label, Multi-center, Dose Escalation Study of GWN323 (Anti-GITR) as a Single Agent and in Combination With PDR001 (Anti-PD-1) in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: Phase I/Ib Study of GWN323 Alone and in Combination With PDR001 in Patients With Advanced Malignancies and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGWN323X2101; 2015-004206-42 (EudraCT Number)
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Solid Tumors; Lymphomas
Keywords: advanced solid tumors; lymphomas; GWN323; PDR001; advanced malignancies; anti-GITR; anti-PD-1; adults
MeSH Terms: conditions — Lymphoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: GWN323
- Arm B (Experimental)
  Interventions: Drug: GWN323; Drug: PDR001

INTERVENTIONS:
Drug: GWN323
Drug: PDR001
  Arms: Arm B

SUMMARY:
The purpose of this trial is to explore the clinical utility of two investigational antibodies in patients with advanced cancer or lymphomas.

This is a multi-center, open-label Phase I/Ib study. The study consists of two dose escalation parts and two dose expansion parts testing GWN323 as a single agent or GWN323 in combination with PDR001. The dose escalation parts will estimate the MTD and/or RDE and test different dosing schedules.

The dose expansion parts of the study will use the MTD/RDE determined in the dose escalation part to assess the activity, safety and tolerability of the investigational products in patients with specific types of cancer and lymphomas.

Approximately 264 adult patients with advanced solid tumors or lymphomas will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic and/or advanced solid tumors or lymphomas not amenable to curative treatment by surgery.
* Histologically documented advanced or metastatic solid tumors or lymphomas
* Must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening
* ECOG Performance Status ≤ 2.

Exclusion Criteria:

* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery).
* Patients diagnosed with T-cell Lymphomas.
* Patients with prior allogenic transplants.
* Patients previously treated with anti-GITR therapy.
* History of severe hypersensitivity reactions to other mAbs.
* Patients intolerant to prior immunotherapy (unable to continue/receive due to immune-related AE).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) - Single Agent | 21 days
  Dose Limiting Toxicities
Incidence of Dose Limiting Toxicities (DLTs) - Combination Agents | 42 days
  Dose Limiting Toxicities

SECONDARY OUTCOMES:
Best Overall Response (BOR), | 36 months
Progression Free Survival (PFS) | 36 months
  per irRC and RECIST v1.1 or Cheson (2014)
Serum concentration profiles of GWN323 as a single agent: Cmax | 36 months
Serum concentration profiles of GWN323 in combination with PDR001 and derived PK parameters: Cmax | 36 months
Presence and titer of anti-GWN323 antibodies | 36 months
Measurement of the effector/regulatory T cell ratio | at screening, 36 months
Serum concentration profiles of GWN323 as a single agent: AUC | 36 months
Serum concentration profiles of GWN323 in combination with PDR001 and derived PK parameters: AUC | 36 months
Presence and titer of anti-PDR001 antibodies | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (4):
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piha-Paul SA, Geva R, Tan TJ, Lim DW, Hierro C, Doi T, Rahma O, Lesokhin A, Luke JJ, Otero J, Nardi L, Singh A, Xyrafas A, Chen X, Mataraza J, Bedard PL. First-in-human phase I/Ib open-label dose-escalation study of GWN323 (anti-GITR) as a single agent and in combination with spartalizumab (anti-PD-1) in patients with advanced solid tumors and lymphomas. J Immunother Cancer. 2021 Aug;9(8):e002863. doi: 10.1136/jitc-2021-002863. PMID 34389618
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17796